CLINICAL TRIAL: NCT03773523
Title: Neuromodulation and Cognitive Training in Opioid Use Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Device Feasibility
Other Study IDs: PSYCH-2018-27116
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Opioid-use Disorder; Opioid Dependence; Opioid Abuse
Keywords: tDCS; Transcranial Direct Current Stimulation; MRI; Opioid dependence; Opioids; Buprenorphine; Suboxone; Lodging Plus; Fairview Lodging Plus
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This study is randomized, double-blind, and sham-controlled. Participants will be randomly assigned to either active or sham tDCS. We are testing device feasibility, safety, and circuit-based targeted engagement.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants will not be informed on their assigned protocol. During consent, they will be informed that there is a 50% chance of being assigned either to the group receiving active tDCS or the group receiving sham tDCS.
  The Principal Investigator and research staff will also be blind to the condition the participant is assigned to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Experimental: active tDCS (Experimental): Subjects that are randomly assigned to this arm will undergo 5 sessions of tDCS.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)
- Sham Comparator: sham tDCS (Sham Comparator): Subjects randomly assigned to sham-tDCS will receive very low current stimulation at the beginning and end of the session, mimicking the feeling of current stimulation in the scalp, but not reaching levels that will stimulate brain function. There will be a total of 5 sham tDCS sessions.
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — tDCS will be performed with Neuroelectrics Starstim Enobio 20, a non-invasive investigational device that has been labeled as a non-significant risk device by the FDA. This study is regulated by the FDA as an Abbreviated IDE. It has built-in safety mechanisms which allow for immediate cessation of stimulation if the subject becomes uncomfortable. The current will be administered via two electrode sponges for 25 mins with 1-2 milliamperes. These administration protocols are in line with protocols that have outlined safe administration (Nitsche 2007; 2008). No side-effects have been reported with the exception of slight itching under the electrode and occasional occurrence of headache, fatigue, or nausea (Poreisz 2007). Electrodes placement: dorsolateral prefrontal cortex (DLPFC); cathode on left DLPFC, anode on right DLPFC.
  Other Names: Starstim

SUMMARY:
The relapsing nature of opioid use disorder is a major obstacle to successful treatment. About 90% of those entering treatment will relapse within one year. To improve treatment outcome, new interventions targeting the underlying brain biomarkers of relapse vulnerability hold significant promise in reducing this critical public health problem. Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique that can modulate brain connectivity.

DETAILED DESCRIPTION:
Cognitive flexibility, the ability to change maladaptive behavior, depends on dorsolateral prefrontal cortex (DLPFC) input to the nucleus accumbens (NAcc; Gruber, Hussain, and O'Donnell 2009). DLPFC stimulation may increase input to NAcc to facilitate proper selection of goal-directed behavior and may also decrease craving in individuals with substance use disorder (Boggio et al. 2008).

We will use transcranial direct current stimulation (tDCS) to stimulate the DLPFC. TDCS is a non-invasive brain stimulation technique that can modulate brain connectivity. TDCS involves applying a weak electrical current (2mA or less) to the scalp via anodal and cathodal electrode sponges, causing either increases or decreases in cortical excitability, respectively. Research has shown in both healthy subjects and patients (e.g. Alzheimer's disease, Parkinson's disease, stroke, and depression) that tDCS has the potential to modulate synaptic strengthening and neurotransmitter-dependent plasticity underlying changes in behavior and learning (Lang et al. 2005).

We are anticipating enrollment of 30 participants. Fifteen participants will be randomly assigned to the interventional tDCS condition, while 15 participants will be randomly assigned to sham tDCS. Both conditions will undergo five sessions of tDCS across five days. Participants will undergo pre- and post-tDCS MRI scans, in addition to clinical interviews and questionnaires. Follow-up interviews will be conducted in person 1 and 2 months after intervention completion to inquire about relapse status.

ELIGIBILITY:
Inclusion Criteria:

* 20 abstinent individuals (18-60 years old; 1-2 weeks of abstinence) who meet DSM-V criteria for opioid use disorder (OUD) will be recruited from the Lodging Plus Program, part of University of Minnesota Medical Center
* This 28-day program provides a supervised environment to treat individuals with OUD in which patients receive random drug screenings. Lodging Plus has 50 beds and admits an average of 20 patients per week and about 50% of patients admitted have a diagnosis of opioid use disorder.
* Ability to provide written consent and comply with study procedures, meet the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) diagnostic criteria for OUD. Subjects may have current comorbid drug use, but their primary substance use disorder diagnosis needs to be based on opioid use. Subjects must have the intention to remain in the Lodging Plus program (4 weeks) until the end of the intervention portion of the study. Vulnerable populations will not be included.

Exclusion Criteria:

* Any medical condition or treatment with neurological sequelae (i.e. stroke, tumor, loss of consciousness>30 min, HIV)
* A head injury resulting in a skull fracture or a loss of consciousness exceeding 30 minutes (i.e., moderate or severe TBI)
* Any contraindications for tDCS or MRI scanning (tDCS contraindication: history of seizures; MRI contraindications; metal implants, pacemakers or any other implanted electrical device, injury with metal, braces, dental implants, non-removable body piercings, pregnancy, breathing or moving disorder)
* DSM-V criteria for psychiatric disorder, may have a lifetime diagnosis of depression
* Presence of a condition that would render study measures difficult or impossible to administer or interpret
* Age outside the range of 18 to 60
* Primary current substance use disorder diagnosis on a substance other than opioid except for caffeine or nicotine
* Clinical evidence for Wernicke-Korsakoff syndrome
* Nicotine use will be recorded.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Change in brain functional connectivity as measured by functional magnetic resonance imaging | Change between baseline and 1-week follow-up
  Investigators will measure magnitude of functional connectivity in between nucleus accumbens (NAcc) and prefrontal cortex (PFC) both at baseline and at follow-up and compare the magnitude of change between the active-tDCS and sham-tDCS groups.

SECONDARY OUTCOMES:
Correlation between functional connectivity change and craving scores | Data collection will be during 2 and 3 weeks of abstinence
  Investigators will (1) compare change in craving scores (difference in craving scores between 2 and 3 weeks of abstinence) between active-tDCS and sham-tDCS groups and (2) conduct parametric correlations between functional connectivity change and change in craving scores.
Correlation between functional connectivity change and clinical outcome | Between 2 weeks of abstinence and 2 months later
  Investigators will record relapse status during the 2 months following treatment discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Jazmin Y Camchong, PhD, Principal Investigator — University of Minnesota; Kelvin O Lim, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Camchong J, Macdonald AW 3rd, Mueller BA, Nelson B, Specker S, Slaymaker V, Lim KO. Changes in resting functional connectivity during abstinence in stimulant use disorder: a preliminary comparison of relapsers and abstainers. Drug Alcohol Depend. 2014 Jun 1;139:145-51. doi: 10.1016/j.drugalcdep.2014.03.024. Epub 2014 Mar 29. PMID 24745476
- [Background] Camchong J, Stenger A, Fein G. Resting-state synchrony during early alcohol abstinence can predict subsequent relapse. Cereb Cortex. 2013 Sep;23(9):2086-99. doi: 10.1093/cercor/bhs190. Epub 2012 Jul 20. PMID 22819968
- [Background] Camchong J, Stenger VA, Fein G. Resting-state synchrony in short-term versus long-term abstinent alcoholics. Alcohol Clin Exp Res. 2013 May;37(5):794-803. doi: 10.1111/acer.12037. Epub 2013 Feb 19. PMID 23421812